CLINICAL TRIAL: NCT00738803
Title: Restoration of Leg Length, Offset, and Center of Rotation in Total Hip Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tennessee Orthopedic Alliance (Other)
Responsible Party: William B Kurtz, Tennessee Orthopedic Alliance
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2615
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Arthritis
Keywords: leg length; hip arthroplasty; offset
MeSH Terms: conditions — Arthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Leg Length and offset measurement arm
  Interventions: Procedure: Total hip replacement

INTERVENTIONS:
Procedure: Total hip replacement — Total hip replacement typically preformed for hip arthritis
  Other Names: Measurement Arm

SUMMARY:
The investigators aim to demonstrate the ability to accurately measure and restore leg length, offset, and center of rotation during a total hip replacement through a new technique that uses the femoral component as a measurement tool. The operative technique requires inserting the femoral component prior to performing the femoral neck osteotomy. After the femoral component is implanted, a reference guide is attached to the femoral component and guides a screw into the ilium at a fixed distance from the femoral component. The pre-arthroplasty measurements of leg length and offset are recorded. The femoral neck osteotomy is performed, and the native femoral head is removed and measured. The acetabular socket is prepared and the acetabular component is inserted. A repeat measurement with trial modular neck components is taken and allows the surgeon an additional opportunity to accurately recreate leg length and offset with the final component. The reference screw is removed from the ilium and the incision is closed.

DETAILED DESCRIPTION:
Background:

Leg length inequality following total hip replacement is the leading cause of patient dissatisfaction and subsequent litigation after total hip replacement. A change in the total offset of the hip (lateral translation of the femur relative to the pelvis) may also cause significant discomfort and hip instability. Before surgery, patients are informed that their leg may be lengthened and a shoe lift may be required in the opposite shoe to equalize the leg lengths. Although much less frequent, the leg can accidentally be shortened following total hip replacement. In one recent study, 62% of patients had a mean leg lengthening of 9 mm and one third of these patients complained about this lengthening.

Limb length inequality can occur for two reasons. First, significant inaccuracies exist in current leg length measurement techniques. Second, the surgeon may deliberately lengthen a patient in order to gain hip stability. Increasing leg length and/or hip offset decreases the occurrence of bony impingement and increases myofascial tension, both of which improve hip stability and prevent hip dislocation.

Current methods of determining leg length and offset during surgery include pre-operative templating, intra-operative measurements, intra-operative x-rays, and computer navigated surgery. From the pre-operative x-rays, surgeons typically determine which size implant will best fit the patient's anatomy and best recreate the same leg length. During surgery, surgeons may attempt to palpate both the operative and the contra-lateral knee and/or ankle to estimate leg lengths. Surgeons may measure the length of the femoral head and neck that were removed and the length of the femoral head and neck that were replaced. Surgeons may insert a long pin into the pelvis (typically the ilium bone) and measure the length from this pin to some reference point on the femur. This pin in the pelvis method is probably considered the most accurate, but the leg must be repositioned in exactly the same position for the measurement to be accurate; 5° of hip abduction results in an 8 mm error in leg length.3 An intra-operative x-ray that shows both hips can also help estimate leg length and hip offset. Surgical navigation can determine leg length but is not widely availability and requires a significant financial commitment by an institution. Surgeons typically determine the appropriate amount of hip offset from their pre-operative templating. Current leg length guides have shown even greater errors in their attempts to measure hip offset.

Hypothesis:

We aim to demonstrate the ability to accurately measure and restore leg length, offset, and center of rotation during a total hip replacement through a new technique that uses the femoral component as a measurement tool. We plan to evaluate the clinical outcome of this procedure and compare it to historical controls.

Goals:

Our primary goal of this research study is to accurately measure and restore the leg length during a hip replacement. Our second goal is to accurately measure and restore the hip offset.

Endpoints:

Patients will be evaluated in clinic at 2 weeks, 3 months, one year, two year, five years and every 5 years afterwards. The leg length, offset and center of rotation will be measured on the pre and post-operative x-ray. Questionnaires based on validated clinical outcomes scores will be completed at the pre-operative visit, at 3 months, one year, two years, five years and every 5 years afterwards.

Abbreviated Methods:

Patients who consent for enrollment in this study will have a standard pre-operative and post-operative AP pelvic x-ray, and leg length, offset measurements, and center of rotation measurements will be made from these two radiographs. In addition, intra-operative fluoroscopic radiographs will also be obtained. Validated questionnaire (Harris Hip Scores) will be administered pre-operatively, at 3 months, at one year, and at two years.

The operative technique for measuring leg length requires inserting the femoral component prior to performing the femoral neck osteotomy. After the femoral component is implanted, a reference guide is attached to the femoral component and guides a screw into the ilium at a fixed distance from the femoral component. The first measurements of leg length and offset are recorded. The reference guide is removed from the femoral component and the femoral neck osteotomy is performed. The native femoral head is removed and measured. The acetabulum is prepared and the acetabular component is inserted. A repeat measurement with trial components in place allows the surgeon an additional opportunity to accurately recreate leg length and offset with the final component. After the final components are inserted, the reference screw is removed from the ilium and the incision is closed. All total hips in this study will be performed through a superior approach so that the anterior and posterior capsules are preserved and hip stability is maximized. This capsular tissue preservation approach will prevent or at least limit the need to deliberately lengthen the leg in order to gain hip stability.

ELIGIBILITY:
Inclusion Criteria:

* Hip arthritis requiring a total hip replacement through a superior approach

Exclusion Criteria:

* Non-english speaking
* Need for a cemented femoral stem
* Acute femoral neck fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Leg Length and total offset | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William B Kurtz, MD, Principal Investigator — Tennessee Orthopedic Alliance
Locations (1):
- Baptist Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Background] Clark CR, Huddleston HD, Schoch EP 3rd, Thomas BJ. Leg-length discrepancy after total hip arthroplasty. J Am Acad Orthop Surg. 2006 Jan;14(1):38-45. doi: 10.5435/00124635-200601000-00007. PMID 16394166
- [Background] Konyves A, Bannister GC. The importance of leg length discrepancy after total hip arthroplasty. J Bone Joint Surg Br. 2005 Feb;87(2):155-7. doi: 10.1302/0301-620x.87b2.14878. PMID 15736733
- [Background] Sarin VK, Pratt WR, Bradley GW. Accurate femur repositioning is critical during intraoperative total hip arthroplasty length and offset assessment. J Arthroplasty. 2005 Oct;20(7):887-91. doi: 10.1016/j.arth.2004.07.001. PMID 16230240